CLINICAL TRIAL: NCT05083949
Title: Relative Bioavailability of Empagliflozin/Metformin Fixed-dose Combination - Empagliflozin 12.5 mg + Metformin 850mg (Boehringer Ingelheim) Coated Tablet Versus Jardiance® 10mg (Reference 1: Boehringer Ingelheim) Coated Tablet and Glifage® 850mg (Reference 2: Merck S / A. ) Coated Tablet, Administered Together in Healthy Male and Female Subjects Under Fed Conditions: an Open-label, Randomised, Single-dose, Two-way Crossover Study
Brief Title: A Study in Healthy Humans to Assess the Relative Bioavailability of One Fixed-dose Combination Tablet Empagliflozin/Metformin Versus Jardiance® Tablet and Glifage® Tablet Administered Together
Acronym: InPedILD®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1276-0041
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2022-09

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Metformin

STUDY DESIGN:
Masking Description: The bioanalytical staff involved are blinded to treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- (A): empagliflozin 10mg (R1)+Glifage® 850mg (R2),then (B): FDC 12.5mg empagliflozin/850mg metformin (Experimental): On Day 1 of Period 1 subjects received treatment A: Single dose tablet of 10 milligram(mg) empagliflozin film-coated and a 850mg of metformin hydrochloride (HCl) (Glifage®) tablet, orally with 200 milliliter(mL) of water.
  On Day 1 of Period 2 subjects received treatment B: Fixed dose combination (FDC) tablet of 12.5mg empagliflozin/850 mg metformin HCl, orally with 200mL of water.
  A high-fat, high-calorie meal was served 30 minutes(min) before drug administration. The treatments were separated by a wash-out phase of at least 7 days.
  Interventions: Drug: FDC 12.5mg empagliflozin/850mg metformin; Drug: Empagliflozin; Drug: Glifage®
- (B): FDC 12.5mg empagliflozin/850mg metformin,then (A): empagliflozin 10mg(R1) + Glifage® 850mg(R2) (Experimental): On Day 1 of Period 1 subjects received treatment B: Fixed dose combination (FDC) tablet containing 12.5 milligram (mg) empagliflozin/850 mg metformin HCl, orally with 200 milliliter (mL) of water.
  On Day 1 of Period 2 subjects received treatment A: Single dose tablet of 10mg empagliflozin and 850 mg of metformin hydrochloride (HCl) (Glifage®) tablet, orally with 200mL of water.
  A high-fat, high-calorie meal was served 30 minutes (min) before drug administration. The treatments were separated by a wash-out phase of at least 7 days.
  Interventions: Drug: FDC 12.5mg empagliflozin/850mg metformin; Drug: Empagliflozin; Drug: Glifage®

INTERVENTIONS:
Drug: FDC 12.5mg empagliflozin/850mg metformin — empagliflozin/metformin
Drug: Empagliflozin — empagliflozin 10mg (R1)
Drug: Glifage® — Glifage® 850mg (R2)
  Other Names: metformin

SUMMARY:
This trial is to establish bioequivalence of the fixed dose combination (FDC) tablets (containing 12.5 mg empagliflozin/850 mg metformin) (Test, T) compared with the single tablets (10 mg empagliflozin and Glifage® 850 mg tablets) (Reference, R).

ELIGIBILITY:
Inclusion criteria:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of at least 18 (inclusive) to 50 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 weight divided by height squared (kg/m2) (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Male subjects, or female subjects who meet any of the following criteria from at least 30 days before the first administration of trial medication until 30 days after trial completion:
* Use of adequate contraception, e.g. any of the following methods plus condom:

  * implants, injectables, combined oral or vaginal contraceptives, intrauterine device
  * Sexually abstinent
  * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
  * Surgically sterilised (including hysterectomy)

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause time from the start of the Q wave to the end of the T wave (QT) / corrected QT (QTc) interval prolongation)
* Smoker (more than 5 cigarettes or 1 cigar or 1 pipe per day)
* Detection or indeterminate / inconclusive result of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) Coronavirus ribonucleic acid (RNA) in the quantitative real-time polymerase chain reaction (RT-qPCR) exam performed on the day before the admission of each period;
* The research participant presents symptoms of coronavirus disease 2019 (COVID-19) infection (even if the result is "undetected" in the RT-PCR exam for COVID-19)
* Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Ciências Farmacêuticas de Estudos e Pesquisas - ICF, Goiânia, Brazil

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to:https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase I, randomised, open label, 2x2 crossover trial in healthy male and female subjects to establish the bioequivalence of 1 Fixed dose combination tablet 12.5 mg empagliflozin/850 mg metformin (treatment B) to the reference treatments (treatment A) which consisted in 1 tablet empagliflozin10 mg (Reference 1) + 1 tablet Glifage® 850 mg (Reference 2).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- (A): Empagliflozin 10mg (R1)+Glifage® 850mg (R2),Then (B): FDC 12.5mg Empagliflozin/850mg Metformin: On Day 1 of Period 1 participants received treatment A: Single dose tablet of 10 milligram(mg) empagliflozin film-coated and a 850mg of metformin hydrochloride (HCl) (Glifage®) tablet, orally with 200 milliliter(mL) of water.
  On Day 1 of Period 2 participants received treatment B: Fixed dose combination (FDC) tablet of 12.5mg empagliflozin/850 mg metformin HCl, orally with 200mL of water.
  A high-fat, high-calorie meal was served 30 minutes(min) before drug administration. The treatments were separated by a wash-out phase of at least 7 days.
- (B): FDC 12.5mg Empagliflozin/850mg Metformin,Then (A): Empagliflozin 10mg(R1) + Glifage® 850mg(R2): On Day 1 of Period 1 participants received treatment B: Fixed dose combination (FDC) tablet containing 12.5 milligram (mg) empagliflozin/850 mg metformin hydrochloride (HCl), orally with 200 milliliter (mL) of water.
  On Day 1 of Period 2 participants received treatment A: Single dose tablet of 10mg empagliflozin and 850 mg of metformin HCl (Glifage®) tablet, orally with 200mL of water.
  A high-fat, high-calorie meal was served 30 minutes (min) before drug administration. The treatments were separated by a wash-out phase of at least 7 days.
Period: Period 1
Arm/Group | (A): Empagliflozin 10mg (R1)+Glifage® 850mg (R2),Then (B): FDC 12.5mg Empagliflozin/850mg Metformin | (B): FDC 12.5mg Empagliflozin/850mg Metformin,Then (A): Empagliflozin 10mg(R1) + Glifage® 850mg(R2)
Started | 16 | 16
Completed | 13 | 14
Not Completed | 3 | 2
Not completed — Positive doping for Tetrahydrocannabinol (THC) | 2 | 1
Not completed — Adverse Event | 1 | 1
Period: Wash-out
Arm/Group | (A): Empagliflozin 10mg (R1)+Glifage® 850mg (R2),Then (B): FDC 12.5mg Empagliflozin/850mg Metformin | (B): FDC 12.5mg Empagliflozin/850mg Metformin,Then (A): Empagliflozin 10mg(R1) + Glifage® 850mg(R2)
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0
Period: Period 2
Arm/Group | (A): Empagliflozin 10mg (R1)+Glifage® 850mg (R2),Then (B): FDC 12.5mg Empagliflozin/850mg Metformin | (B): FDC 12.5mg Empagliflozin/850mg Metformin,Then (A): Empagliflozin 10mg(R1) + Glifage® 850mg(R2)
Started | 13 | 14
Completed | 12 | 12
Not Completed | 1 | 2
Not completed — The patient was not able to eat the full content of the breakfast | 1 | 0
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The treated set included all participants in the research that were randomized and treated with at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | (A): Empagliflozin 10mg (R1)+Glifage® 850mg (R2),Then (B): FDC 12.5mg Empagliflozin/850mg Metformin | (B): FDC 12.5mg Empagliflozin/850mg Metformin,Then (A): Empagliflozin 10mg(R1) + Glifage® 850mg(R2) | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.0 (7.2) | 31.7 (8.3) | 31.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 7 | 11 | 18
  More than one race | 6 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Dose-normalized Area Under the Concentration-time Curve of Empagliflozin in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of empagliflozin in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) normalized to the actual administered dose is presented. The AUC0-tz was divided by the actual dose strength to get the normalized area under the concentration-time curve. The statistical model used for the analysis of the primary endpoints was an analysis of variance (ANOVA) on the logarithmic scale. That is, the PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: sequence, subjects within sequences, period and treatment. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed. Unit of measure:(hour*nanogram/milliliter)/milligram.
Time Frame: Within 5 minutes (min) before and 15min, 30min, 45min, 1h, 1h15min, 1h30min, 1h45min, 2h, 2h20min, 2h40min, 3h, 3h30min, 4h, 4h30min, 5h, 5h30min, 6h, 7h, 8h, 10h, 12h, 24h, 48h, and 72h after treatment administration for both arms.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This set included all subjects who provided all PK endpoints for all treatment periods that were defined as primary (Cmax and AUCo-tz) and was not excluded due to a protocol violation relevant to the evaluation of PK or due to PK non-evaluability. Only subjects with non-missing values were included.
Measure: Geometric Least Squares Mean (Standard Error); unit: (h*ng/mL)/mg
Groups:
- (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2): Participants received treatment A: Single dose tablet of 10 milligram (mg) empagliflozin film-coated and a 850mg of metformin HCl (Glifage®) tablet, orally with 200 milliliter (mL) of water.
  A high-fat, high-calorie meal was served 30 minutes (min) before drug administration.
- (B): FDC 12.5mg Empagliflozin/850mg Metformin: Participants were administered the treatment B which consisted of a single Fixed dose combination (FDC) tablet containing 12.5 milligram (mg) empagliflozin/850 mg metformin HCl, orally with 200 milliliter (mL) of water. A high-fat, high-calorie meal was served 30 minutes (min) before drug administration.
Arm/Group | (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) | (B): FDC 12.5mg Empagliflozin/850mg Metformin
Number analyzed (Participants) | 24 | 24
(h*ng/mL)/mg | 117.15 (NA) — The standard error is actually the geometric standard error and is equal to 1.04. | 116.65 (NA) — The standard error is actually the geometric standard error and is equal to 1.04.
Statistical Analysis 1: Comparison: (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) vs (B): FDC 12.5mg Empagliflozin/850mg Metformin; The statistical model used for the analysis was an analysis of variance (ANOVA) on the logarithmic scale. That is, the PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: sequence, subjects within sequences, period and treatment. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; Test type: Equivalence — Bioequivalence was concluded, if the confidence interval (CI) for the comparison of geometric least squares means ratio was included in the pre-defined equivalence range of 80.00% to 125.00%; p = 0.7792, ANOVA; Ratio of GLSM (%) = 99.57, 90% CI 2-sided [97.03 to 102.19], Standard Deviation 5.23 — Ratio of Geometric Least Squares Means (GLSM) was calculated as: Fixed dose combination (treatment B)/ free dose combination (treatment A). Standard deviation is actually intra-individual geometric coefficient of variation (gCV [%])

2. Primary Outcome: Dose-normalized Maximum Measured Concentration of Empagliflozin (Cmax)
Description: Dose-normalized Maximum measured concentration of empagliflozin in plasma is presented. The maximum measured concentration was divided by the actual dose strength to get the dose-normalised Cmax. The statistical model used for the analysis of the primary endpoints was an analysis of variance (ANOVA) on the logarithmic scale. That is, the PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: sequence, subjects within sequences, period and treatment. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed. The unit of measure reported is: (nanogram/milliliter)/milligram.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: (ng/mL)/mg
Arm/Group | (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) | (B): FDC 12.5mg Empagliflozin/850mg Metformin
Number analyzed (Participants) | 24 | 24
(ng/mL)/mg | 13.42 (NA) — The standard error is actually the geometric standard error and is equal to 1.03. | 13.60 (NA) — The standard error is actually the geometric standard error and is equal to 1.03.
Statistical Analysis 1: Comparison: (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) vs (B): FDC 12.5mg Empagliflozin/850mg Metformin; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.6493, ANOVA; Ratio of GLSM (%) = 101.36, 90% CI 2-sided [96.39 to 106.59], Standard Deviation 10.18 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Area Under the Concentration-time Curve of Metformin in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of metformin in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is presented. The statistical model used for the analysis of the primary endpoints was an analysis of variance (ANOVA) on the logarithmic scale. That is, the PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: sequence, subjects within sequences, period and treatment. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed.
Time Frame: Within 5 minutes(min) before and 15min, 30min, 45min, 1h, 1h15min, 1h30min, 1h45min, 2h, 2h20min, 2h40min, 3h, 3h30min, 4h, 4h30min, 5h, 5h30min, 6h, 7h, 8h, 10h, 12h, 24h, 48h, and 72h after treatment administration for both arms.
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanogram/milliliter (h*ng/mL)
Arm/Group | (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) | (B): FDC 12.5mg Empagliflozin/850mg Metformin
Number analyzed (Participants) | 24 | 24
hour*nanogram/milliliter (h*ng/mL) | 10299.45 (NA) — The standard error is actually the geometric standard error and is equal to 1.05. | 10467.41 (NA) — The standard error is actually the geometric standard error and is equal to 1.05.
Statistical Analysis 1: Comparison: (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) vs (B): FDC 12.5mg Empagliflozin/850mg Metformin; The statistical model used for the analysis of the was an analysis of variance (ANOVA) on the logarithmic scale. That is, the PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: sequence, subjects within sequences, period and treatment. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.4710, ANOVA; Ratio of GLSM (%) = 101.63, 90% CI 2-sided [97.85 to 105.55], Standard Deviation 7.65 — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Maximum Measured Concentration of Metformin (Cmax)
Description: Maximum measured concentration of metformin in plasma is presented. The statistical model used for the analysis of the primary endpoints was an analysis of variance (ANOVA) on the logarithmic scale. That is, the PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: sequence, subjects within sequences, period and treatment. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanogram/milliliter (ng/mL )
Arm/Group | (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) | (B): FDC 12.5mg Empagliflozin/850mg Metformin
Number analyzed (Participants) | 24 | 24
nanogram/milliliter (ng/mL ) | 1333.58 (NA) — The standard error is actually the geometric standard error and is equal to 1.04. | 1308.39 (NA) — The standard error is actually the geometric standard error and is equal to 1.04.
Statistical Analysis 1: Comparison: (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) vs (B): FDC 12.5mg Empagliflozin/850mg Metformin; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.4251, ANOVA; Ratio of GLSM (%) = 98.11, 90% CI 2-sided [94.24 to 102.15], Standard Deviation 8.14 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Dose-normalized Area Under the Concentration-time Curve of Empagliflozin in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞ )
Description: Area under the concentration-time curve of empagliflozin in plasma over the time interval from 0 extrapolated to infinity from the last quantifiable data point (AUC0-inf) normalized to the actual administered dose is presented. The AUC0-oo was divided by the actual dose strength to get the normalized area under the concentration-time curve. The statistical model used for the analysis of the primary endpoints was an analysis of variance (ANOVA) on the logarithmic scale. That is, the PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: sequence, subjects within sequences, period and treatment. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed. Unit of measure: (hour*nanogram/milliliter)/milligram.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: (h*ng/mL)/mg
Groups:
- (B):FDC 12.5mg Empagliflozin/850mg Metformin: Participants were administered the treatment B which consisted of a single Fixed dose combination (FDC) tablet containing 12.5 milligram (mg) empagliflozin/850 mg metformin HCl, orally with 200 milliliter (mL) of water. A high-fat, high-calorie meal was served 30 minutes (min) before drug administration.
Arm/Group | (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) | (B):FDC 12.5mg Empagliflozin/850mg Metformin
Number analyzed (Participants) | 24 | 24
(h*ng/mL)/mg | 118.25 (NA) — The standard error is actually the geometric standard error and is equal to 1.03. | 117.64 (NA) — The standard error is actually the geometric standard error and is equal to 1.03.
Statistical Analysis 1: Comparison: (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) vs (B):FDC 12.5mg Empagliflozin/850mg Metformin; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.7379, ANOVA; Ratio of GLSM (%) = 99.49, 90% CI 2-sided [96.93 to 102.11], Standard Deviation 5.25 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Area Under the Concentration-time Curve of Metformin in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of metformin in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞ ) is presented. The statistical model used for the analysis was an analysis of variance (ANOVA) on the logarithmic scale. That is, the PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. This model included effects accounting for the following sources of variation: sequence, subjects within sequences, period and treatment. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanogram/milliliter (hr*ng/mL)
Arm/Group | (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) | (B): FDC 12.5mg Empagliflozin/850mg Metformin
Number analyzed (Participants) | 24 | 24
hour*nanogram/milliliter (hr*ng/mL) | 10440.79 (NA) — The standard error is actually the geometric standard error and is equal to 1.05. | 10570.45 (NA) — The standard error is actually the geometric standard error and is equal to 1.05.
Statistical Analysis 1: Comparison: (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) vs (B): FDC 12.5mg Empagliflozin/850mg Metformin; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.5895, ANOVA; Ratio of GLSM (%) = 101.24, 90% CI 2-sided [97.40 to 105.24], Standard Deviation 7.82 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Time From Last Dosing to the Maximum Measured Concentration of Empagliflozin in Plasma (Tmax)
Description: Time from last dosing to the maximum measured concentration of empagliflozin in plasma (tmax) is presented.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours (hr)
Arm/Group | (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) | (B): FDC 12.5mg Empagliflozin/850mg Metformin
Number analyzed (Participants) | 24 | 24
Hours (hr) | 2.33 [1.25 to 5.00] | 2.17 [1.00 to 5.50]

8. Secondary Outcome: Time From Last Dosing to the Maximum Measured Concentration of Metformin in Plasma (Tmax)
Description: Time from last dosing to the maximum measured concentration of metformin in plasma (tmax) is presented.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours (hr)
Arm/Group | (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) | (B): FDC 12.5mg Empagliflozin/850mg Metformin
Number analyzed (Participants) | 24 | 24
Hours (hr) | 4.00 [3.00 to 4.50] | 4.00 [1.00 to 5.00]

9. Secondary Outcome: Percentage (%) of the AUC of Empagliflozin That Has Been Derived After Extrapolation
Description: The percentage (%) of the AUC of empagliflozin that has been derived after extrapolation is reported.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) | (B): FDC 12.5mg Empagliflozin/850mg Metformin
Number analyzed (Participants) | 24 | 24
Percentage (%) | 9.77 (3.04) | 9.31 (1.87)

10. Secondary Outcome: Percentage (%) of the AUC of Metformin That Has Been Derived After Extrapolation
Description: The percentage (%) of the AUC of metformin that has been derived after extrapolation is reported.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) | (B): FDC 12.5mg Empagliflozin/850mg Metformin
Number analyzed (Participants) | 24 | 24
Percentage (%) | 14.35 (8.50) | 13.04 (5.58)

11. Secondary Outcome: Terminal Half-life of Empagliflozin in Plasma (t1/2)
Description: The terminal half-life of empagliflozin in plasma (t1/2) is presented.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours (hr)
Groups:
- (A): Empaglifozin 10mg (R1) + Metformin (Glifage®) 850mg (R2): Participants received treatment A: Single dose tablet of 10 milligram (mg) empagliflozin film-coated and a 850mg of metformin HCl (Glifage®) tablet, orally with 200 milliliter (mL) of water.
  A high-fat, high-calorie meal was served 30 minutes (min) before drug administration.
Arm/Group | (A): Empaglifozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) | (B): FDC 12.5mg Empagliflozin/850mg Metformin
Number analyzed (Participants) | 24 | 24
Hours (hr) | 0.08 [0.04 to 0.11] | 0.08 [0.05 to 0.11]

12. Secondary Outcome: Terminal Half-life of Metformin in Plasma (t1/2)
Description: The terminal half-life of metformin in plasma (t1/2) is presented.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours (hr)
Arm/Group | (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) | (B): FDC 12.5mg Empagliflozin/850mg Metformin
Number analyzed (Participants) | 24 | 24
Hours (hr) | 0.06 [0.02 to 0.13] | 0.06 [0.02 to 0.11]

13. Secondary Outcome: Elimination Rate Constant (Kel) for Empagliflozin
Description: The elimination rate constant (Kel) for empagliflozin is reported.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hours (1/hr)
Arm/Group | (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) | (B): FDC 12.5mg Empagliflozin/850mg Metformin
Number analyzed (Participants) | 24 | 24
1/hours (1/hr) | 0.93 (0.61) | 0.84 (0.44)

14. Secondary Outcome: Elimination Rate Constant (Kel) for Metformin
Description: The elimination rate constant (Kel) for metformin is reported.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hours (1/hr)
Arm/Group | (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) | (B): FDC 12.5mg Empagliflozin/850mg Metformin
Number analyzed (Participants) | 24 | 24
1/hours (1/hr) | 1.33 (2.14) | 0.97 (1.02)

ADVERSE EVENTS:
Time Frame: Up to 14 days after the last treatment administration.
Description: Treated Set (TS): The treated set included all participants in the research that were randomized and treated with at least one dose of study medication.
Arm/Group | (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) | (B): FDC 12.5mg Empagliflozin/850mg Metformin
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 5/30 | 2/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | (A): Empagliflozin 10mg (R1) + Metformin (Glifage®) 850mg (R2) (N=30) | (B): FDC 12.5mg Empagliflozin/850mg Metformin (N=29)
White blood cells in urine (Investigations) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT05083949/Prot_SAP_000.pdf